CLINICAL TRIAL: NCT04706845
Title: Understanding the Burden of ACC Through the Eyes of Patients
Status: Completed | Type: Observational
Sponsor: Ayala Pharmaceuticals, Inc, (Industry)
Collaborators: Adenoid Cystic Carcinoma Research Foundation (Other); Memorial Sloan Kettering Cancer Center (Other); Hadassah Medical Organization (Other); Engage Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL Patient Burden 01
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: No evident disease
- 2: Metastatic Disease; Watchful Waiting: Tumors bearing NOTCH Mutation
- 3: Metastatic Disease; Watchful Waiting: Tumors bearing Notch Wild Type
- 4: Progressive Disease: Tumors bearing NOTCH Mutation
- 5: Progressive Disease: Tumors bearing Notch Wild Type

SUMMARY:
This is a comprehensive, cross-sectional study conducted with approximately 40-60 individuals affected by ACC who may know the results of molecular profiling of their tumor.

Primary Objectives:

* To identify the specific burdens faced by patients with ACC
* To compare/contrast the burdens faced by patients with ACC at different disease stages (no evident disease, metastatic disease/watchful waiting, progressive disease)

DETAILED DESCRIPTION:
This is a comprehensive, cross-sectional study conducted with approximately 40-60 individuals affected by ACC who may know the results of molecular profiling of their tumor.

Primary Objectives:

* To identify the specific burdens faced by patients with ACC
* To compare/contrast the burdens faced by patients with ACC at different disease stages (no evident disease, metastatic disease/watchful waiting, progressive disease)

Secondary Objectives:

* To assess QoL implication in patients living with ACC (Adenoid Cystic Carcinoma)
* To compare the burdens and QoL impacts in people living with ACC, with their tumors bearing Notch mutations or Notch Wild Type due to:

  * Rate of disease progression
  * Location of Metastases

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a person diagnosed with ACC who is 18 years or older
2. For patients with metastatic disease; watchful waiting or progressive disease, participants must know the results of molecular profiling of their tumor
3. Histologically-confirmed diagnosis of ACC with written proof of disease and molecular profile of tumor provided. This can be a note showing genetic diagnosis from a relevant testing laboratory, physician consult notes, a medical record of diagnosis, or any other single piece of documentation that connects your name/the patient's name with ACC.
4. Able to read, write and understand English, Hebrew, Arabic, or Russian
5. Able to grant informed consent
6. Willing to participate in a 45-to-60-minute telephone interview, including follow up questions (if necessary)

Exclusion Criteria:

1. Inability to meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within the United States or Israel, patients who have been diagnosed with Adenoid Cystic Carcinoma (ACC)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Key burdens related to the disease or treatments | Q4-2021
Life impacts of those burdens for patient/family | Q4-2021

CONTACTS AND LOCATIONS:
Locations (1):
- Engage Health, Eagan, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No